CLINICAL TRIAL: NCT02457975
Title: Near-Infrared Photobiomodulation for the Treatment of Diabetic Macular Edema
Brief Title: Photobiomodulation for the Treatment of Diabetic Macular Edema
Acronym: PTDME
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Judy Kim, Professor of Ophthalmology, Medical College of Wisconsin
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00024065
Record Dates: First submitted 2015-05-25; First posted 2015-05-29 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Macular Edema; Photobiomodulation; Phototherapy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — aflibercept; Bevacizumab; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravitreous VEGF-inhibitors (Active Comparator): Three intravitreous VEGF inhibitors - aflibercept (Eylea, Regeneron Pharmaceuticals), bevacizumab (Avastin, Genentech), and ranibizumab (Lucentis, Genentech) - are commonly used for the treatment of diabetic macular edema causing vision impairment and have been shown to be beneficial and relatively safe. Study participants in the anti-VEGF group will be treated with intravitreous injections of one of these agents: afibercept (2.0 mg), bevacizumab (1.25 mg) or ranibizumab (0.5 mg) at appropriate intervals as determined by the treating ophthalmologist.
  Interventions: Drug: intravitreous VEGF-inhibitors
- 670nm PBM plus VEGF-inhibitors (Experimental): Subjects in the 670 nm Photobiomodulation (PBM) intervention arm will be treated (in addition to Anti-VEGF treatment) with 670nm light (WARP10, Quantum, Devices, Inc, Barneveld, WI). The portable, battery-operated 670 nm LED array specifically designed not to generate heat will be held 1 inch from the closed treatment eye. A 90-sec light treatment will be delivered. After 90 sec a timer turns off the light. The dose of light delivered at the surface of the cornea is calculated to be 4.5 J/cm2 (90 sec x 0.05 W/cm2 = 4.5 J/cm2). PBM treatment will be applied for 90 sec once per day, three consecutive days per week for 8 weeks. Previous clinical studies, have shown this treatment regimen and dose to be safe and effective in the treatment of dry AMD and non-center involving DME
  Interventions: Device: 670nm PBM; Drug: intravitreous VEGF-inhibitors

INTERVENTIONS:
Device: 670nm PBM — Battery operated, hand-held, 10 cm2 Light Emitting Diode (LED) array designed to deliver 50 mW/cm2 of light for 90 seconds resulting in a light dose of 4.5 Joules/cm2
  Other Names: WARP10 by Quantum Devices, Inc (Barneveld, WI)
  Arms: 670nm PBM plus VEGF-inhibitors
Drug: intravitreous VEGF-inhibitors — Threeintravitreous VEGF inhibitors - aflibercept (Eylea, Regeneron Pharmaceuticals), bevacizumab (Avastin, Genentech), and ranibizumab (Lucentis, Genentech) - are commonly used for the treatment of diabetic macular edema causing vision impairment and have been shown to be beneficial and relatively safe. Study participants in the anti-VEGF group will be treated with intravitreous injections of one of these agents: afibercept (2.0 mg), bevacizumab (1.25 mg) or ranibizumab (0.5 mg) at appropriate intervals as determined by the treating ophthalmologist.
  Other Names: aflibercept, bevacizumab, or ranibizumab

SUMMARY:
The current application proposes to conduct a prospective, clinical trial in diabetic subjects with diabetic macular edema (DME) to evaluate the therapeutic efficacy of 670 nm photobiomodulation on validated clinical outcome measures and anatomical changes in central macula by optical coherence tomography (OCT) and other imaging modalities. A total of 30 diabetic patients with treatment-refractory clinically significant diabetic macular edema will be included in this study and randomized into two equal groups. One eye per participant will be included to avoid exposure of both eyes to the study intervention. If both eyes are eligible, the eye with worse visual acuity will become the study eye. One group will be treated with standard-of-care (intravitreal anti-VEGF agent) injections. The photobiomodulaton (PBM) intervention group will be treated with the standard-of-care intravitreal anti-VEGF (vascular endothelial growth factor) injections and 670 nm PBM in one eye. Baseline functional and anatomic assessments will be made and anti-VEGF therapy will be administered as determined by the treating Ophthalmologist.

DETAILED DESCRIPTION:
A total of 30 diabetic patients with treatment-refractory clinically significant diabetic macular edema will be included in this study and randomized into two equal groups. One eye per participant will be included to avoid exposure of both eyes to the study intervention. If both eyes are eligible, the eye with worse visual acuity will become the study eye. One group will be treated with standard-of-care (intravitreal anti-VEGF agent) injections. The PBM intervention group will be treated with the standard-of-care intravitreal anti-VEGF injections and 670 nm PBM in one eye. Baseline functional and anatomic assessments will be made and anti-VEGF therapy will be administered as determined by the treating Ophthalmologist.

Subjects in the PBM intervention arm will be treated (in addition to standard care) with 670nm light (WARP10, Quantum, Devices, Inc, Barneveld, WI). The portable, battery-operated 670 nm LED array specifically designed not to generate heat will be hand held 1 inch from the closed treatment eye. An 80-sec light treatment will be delivered. After 80 sec a timer turns off the light. The dose of light delivered at the surface of the cornea is calculated to be 4.0 J/cm2 (80 sec x 0.05 W/cm2 = 4.0 J/cm2). PBM treatment will be applied for 80 sec once per day, three consecutive days per week for 8 weeks. Previous clinical studies, have shown this treatment regimen and dose to be safe and effective in the treatment of dry AMD and non-center involving DME.

ASSESSMENTS: Subjects will undergo a detailed functional and structural evaluation at baseline and at 8 and 24 weeks. Seven-field color fundus photographs will be obtained for ETDRS retinopathy grading at baseline 8 and 24 weeks. Best corrected visual acuity (BCVA) Early Treatment Diabetic Retinopathy Study (ETDRS) will be obtained at every visit. Fundus fluorescein angiography and Spectralis OCT scans will be obtained according to predefined protocols. Blood pressure and glycosylated hemoglobin level will be recorded at baseline and 8 and 24 weeks to identify any changes in systemic status that could affect retinopathy grade and macular edema. Cataract status will be recorded at baseline and 8 and 24 weeks as a safety measure and as a possible confounding factor for visual acuity assessment.

OUTCOME MEASURES: Functional measure will be change in ETDRS BCVA from baseline. Structural outcome measures will include changes in qualitative and quantitative OCT parameters, including macular thickness and volume in 9 ETDRS subfields, obtained from automated measures in the Heidelberg Eye Explorer software (Heidelberg Engineering GmbH, Heidelberg, Germany) without formally correcting for boundary detection error; these measures are highly reproducible. Changes in intraretinal and subretinal fluid on OCT will be evaluated. The change in ETDRS severity grade of diabetic retinopathy will be reported from 7-field color fundus photographs. Safety parameters will include the reporting of ocular and nonocular adverse events. Changes to the greatest linear dimension and area of the foveal avascular zone on fluorescein angiography, together with the degree of perifoveal capillary loss, will be reported. The grading of photographs both for retinopathy grade and foveal avascular zone measurements will be carried out by a trained and certified senior diabetic retinopathy grader at the Medical College of Wisconsin. The number of anti-VEGF treatments in the two arms will be compared as a secondary measure of effect of PBM.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with type 1 or 2 diabetes

Exclusion Criteria:

Uncontrolled glaucoma; aphasia cataract precluding fundus photography; external ocular infections; previous anti-VEGF or laser treatment in the preceding 3 months in both eyes; angiographic evidence of macular ischemia macular edema glycosylated hemoglobin of more than 11.0% past medical history of chronic renal failure an arteriothrombotic event within 6 months before randomization pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Visual Acuity as assessed by the Early Treatment of Diabetic Retinopathy Study (EDTRS) Classification | Change from baseline at 8 weeks; Change from baseline at 24 weeks

SECONDARY OUTCOMES:
Spectral Density-Optical Coherence Tomography (SD-OCT) | Change from baseline at 8 weeks; Change from baseline at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Judy Kim, MD, Principal Investigator — MCW Dept of Ophthalmology; Sandeep Gopalakrishnan, Ph.D., Principal Investigator — UW-Milwaukee
Locations (1):
- Medical College of Wisconsin Froedert Hospital, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Zhang X, Zeng H, Bao S, Wang N, Gillies MC. Diabetic macular edema: new concepts in patho-physiology and treatment. Cell Biosci. 2014 May 14;4:27. doi: 10.1186/2045-3701-4-27. eCollection 2014. PMID 24955234
- [Background] Falavarjani KG, Nguyen QD. Adverse events and complications associated with intravitreal injection of anti-VEGF agents: a review of literature. Eye (Lond). 2013 Jul;27(7):787-94. doi: 10.1038/eye.2013.107. Epub 2013 May 31. PMID 23722722
- [Background] Tang J, Herda AA, Kern TS. Photobiomodulation in the treatment of patients with non-center-involving diabetic macular oedema. Br J Ophthalmol. 2014 Aug;98(8):1013-5. doi: 10.1136/bjophthalmol-2013-304477. Epub 2014 Mar 28. PMID 24682183
- [Background] Simo R, Sundstrom JM, Antonetti DA. Ocular Anti-VEGF therapy for diabetic retinopathy: the role of VEGF in the pathogenesis of diabetic retinopathy. Diabetes Care. 2014 Apr;37(4):893-9. doi: 10.2337/dc13-2002. PMID 24652720
- [Background] Eells JT, Wong-Riley MT, VerHoeve J, Henry M, Buchman EV, Kane MP, Gould LJ, Das R, Jett M, Hodgson BD, Margolis D, Whelan HT. Mitochondrial signal transduction in accelerated wound and retinal healing by near-infrared light therapy. Mitochondrion. 2004 Sep;4(5-6):559-67. doi: 10.1016/j.mito.2004.07.033. PMID 16120414
- [Background] Tang J, Du Y, Lee CA, Talahalli R, Eells JT, Kern TS. Low-intensity far-red light inhibits early lesions that contribute to diabetic retinopathy: in vivo and in vitro. Invest Ophthalmol Vis Sci. 2013 May 1;54(5):3681-90. doi: 10.1167/iovs.12-11018. PMID 23557732
- [Background] Cheung N, Wong IY, Wong TY. Ocular anti-VEGF therapy for diabetic retinopathy: overview of clinical efficacy and evolving applications. Diabetes Care. 2014 Apr;37(4):900-5. doi: 10.2337/dc13-1990. PMID 24652721
- [Background] Eells JT, Henry MM, Summerfelt P, Wong-Riley MT, Buchmann EV, Kane M, Whelan NT, Whelan HT. Therapeutic photobiomodulation for methanol-induced retinal toxicity. Proc Natl Acad Sci U S A. 2003 Mar 18;100(6):3439-44. doi: 10.1073/pnas.0534746100. Epub 2003 Mar 7. PMID 12626762
- [Background] Chung H, Dai T, Sharma SK, Huang YY, Carroll JD, Hamblin MR. The nuts and bolts of low-level laser (light) therapy. Ann Biomed Eng. 2012 Feb;40(2):516-33. doi: 10.1007/s10439-011-0454-7. Epub 2011 Nov 2. PMID 22045511
- See also: TORPA Study of Photobiomdulation for AMD — http://clinicaltrials.gov/ct2/show/NCT00940407